CLINICAL TRIAL: NCT06900543
Title: A Randomized, Open-label, Multicenter Study Comparing the Efficacy and Safety of NRT6003 Injection With Conventional Transarterial Chemoembolization (cTACE) in Chinese Patients With Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: Chinese HCC Efficacy Evaluation, Response and Safety Study of TareSphere
Acronym: CHEERS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu New Radiomedicine Technology Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRT6003-HCC-2024; CTR20250792 (Other: Center for Drug Evaluation, NMPA)
Record Dates: First submitted 2025-03-17; First posted 2025-03-28 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Selective internal radiation therapy; Yttrium-90; Transarterial Radioembolization; Conventional Transarterial Chemoembolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NRT6003 Injection (Experimental): Selective internal radiation therapy (SIRT) with TareSphere
  Interventions: Drug: NRT6003 Injection
- cTACE (Active Comparator): Transarterial chemoembolization
  Interventions: Drug: cTACE

INTERVENTIONS:
Drug: NRT6003 Injection — Patients will be administered NRT6003 Injection via Intra-arterial infusion, and subsequently they will be assessed by PET/CT imaging within 24 hours for its distribution in the chest and upper abdomen, including extrahepatic shunts, intrahepatic distribution, and target lesion distribution as expected.
  Other Names: Yttrium-90 carbon microspheres
  Arms: NRT6003 Injection
Drug: cTACE — Patients will receive cTACE treatment. And the investigators will select one or more chemotherapy drugs in combination with embolic materials for administration, based on the specific condition of the patient.
  Other Names: transarterial chemoembolization
  Arms: cTACE

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of NRT6003 Injection compared to cTACE in patients with unresectable HCC.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

1. Does NRT6003 Injection improve tumor response rates compared to cTACE in patients with unresectable HCC?
2. What adverse events do participants experience when receiving NRT6003 Injection compared to cTACE?

Investigators will compare NRT6003 Injection to cTACE to determine:

1. Whether NRT6003 Injection demonstrates superior efficacy in tumor control and long-term survival (e.g., objective response rate, time to progression, etc.).
2. Whether NRT6003 Injection has a comparable or improved safety profile vs. cTACE (e.g., incidence of adverse events, etc.).

Participants will:

1. Receive either NRT6003 Injection or cTACE as per randomized assignment.
2. Undergo scheduled follow-up visits for imaging assessments (e.g., MRI or CT scans, etc.) and safety evaluations.
3. Provide blood samples for biomarker analysis.
4. Report any symptoms or medical events through a patient diary and during clinic visits.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosed as hepatocellular carcinoma (CNLC Ⅰa-Ⅲa) clinically, by imaging and/or pathology based on the guideline of the National Health Commission of the People's Republic of China (2024).
2. Evaluated by the investigator as not suitable for surgical resection/ablation/liver transplantation, or there is high risk for surgical resection, or the participant refuses surgical resection/ablation/liver transplantation.
3. Child-Pugh score ≤ 7.
4. Eastern Cooperative Oncology Group performance status ≤ 1.
5. Adequate organ function.

Key Exclusion Criteria:

1. Imaging evidence or suspicion of extrahepatic metastases (including regional lymph node metastases).
2. Prior antitumor treatment for primary hepatocellular carcinoma.
3. Prior external radiation therapy or intra-arterial brachytherapy.
4. Liver vascular evaluation results that do not meet all the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time to Progression (TTP) | Through study completion, at least 18 months
  Evaluated by the Blinded Independent Review Committee (BIRC) in accordance with the mRECIST criteria

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, at least 18 months
  Evaluated by the Blinded Independent Review Committee (BIRC) in accordance with the mRECIST criteria
Duration of Response (DOR) | Through study completion, at least 18 months
  Evaluated by the Blinded Independent Review Committee (BIRC) in accordance with the mRECIST criteria
Localized Time to Progression (localized TTP) | Through study completion, at least 18 months
  Evaluated by the Blinded Independent Review Committee (BIRC) in accordance with the mRECIST criteria
Time to Progression | Through study completion, at least 18 months
  Evaluated by the investigator in accordance with the mRECIST criteria
Localized Time to Progression | Through study completion, at least 18 months
  Evaluated by the investigator in accordance with the mRECIST criteria
Objective Response Rate | Through study completion, at least 18 months
  Evaluated by the investigator in accordance with the mRECIST criteria
Duration of Response | Through study completion, at least 18 months
  Evaluated by the investigator in accordance with the mRECIST criteria
Surgery Rate | From the administration to study completion, at least 18 months
  Resection rate of liver target lesions
Overall Survival (OS) | From the administration to study completion, at least 18 months
  Based on survival follow-up information
Changes in Tumor Biomarkers | From the administration to study completion, at least 18 months
  The variation of alpha fetoprotein (AFP) levels
Incidence and severity of adverse events (AE) and severe adverse events (SAE) | Throughout the study, at least 18 months
  In accordance with NCI-CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Teng, Principal Investigator — Zhongda Hospital
Locations (11):
- China (11):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - West China Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No